CLINICAL TRIAL: NCT02939313
Title: Charleston ARC Clinical Project 4 Cortical rTMS as a Tool to Change Craving and Brain Reactivity to Alcohol Cues
Brief Title: Cortical rTMS as a Tool to Change Brain Reactivity to Alcohol Cues
Acronym: ARC4
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 00050256; P50AA010761 (NIH); NCT02948296 (obsolete NCT alias)
Record Dates: First submitted 2016-09-01; First posted 2016-10-20 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Alcohol Dependance
Keywords: alcohol; addiction; cTBS
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- medial prefrontal (Experimental): Individuals will receive medial prefrontal cortex stimulation
  Interventions: Device: medial prefrontal cortex
- dorsolateral prefrontal (Experimental): Individuals will receive dorsolateral prefrontal cortex stimulation
  Interventions: Device: dorsolateral prefrontal cortex
- sham (Sham Comparator): Individuals will receive sham stimulation to the medial prefrontal and dorsolateral prefrontal cortex
  Interventions: Device: sham

INTERVENTIONS:
Device: medial prefrontal cortex — a form of theta burst stimulation that noninvasively induces a depression in brain reactivity
  Other Names: medial prefrontal
  Arms: medial prefrontal
Device: dorsolateral prefrontal cortex — a form of transcranial magnetic stimulation that noninvasively induces an increase in brain reactivity
  Other Names: dorsolateral prefrontal
  Arms: dorsolateral prefrontal
Device: sham — sham stimulation
  Arms: sham

SUMMARY:
The goal of this investigation is to determine if, in heavy alcohol users, a single session of transcranial magnetic brain stimulation (TMS) over a brain region involved in craving (medial prefrontal cortex) and a brain region involved in cogntive control (dorsolateral prefrontal cortex) can lower an individual's craving and brain response to alcohol cues. This study involves a screening visit, followed by three visits which involve brain imaging (using functional MRI) and brain stimulation (using TMS). There is also an additional Magnetic resonance spectroscopy (MRS) exploratory Aim in which we will measure the concentration of glutamate in the prefrontal cortex before and after a session of TMS.

DETAILED DESCRIPTION:
Alcohol Use Disorders (AUDs) are prevalent, devastating, and difficult to treat. High relapse rates are likely due to factors that affect limbic and executive circuits in the brain, including vulnerability to salient cues and loss of cognitive control. Limbic drive and executive control are regulated by two cortical-subcortical neural circuits -the limbic loop that includes projections from the medial prefrontal cortex (mPFC) to the ventral striatum, and the executive control loop that includes projections from the dorsolateral prefrontal cortex (dlPFC) to the dorsal striatum. Optogenetic manipulation in animals has demonstrated a causal relationship between activity in these frontal-striatal circuits and drinking behavior. Consequently, an innovative and potentially fruitful new strategy in the treatment of AUDs in humans would be to selectively attenuate limbic circuitry (to reduce reward salience), and/or amplify executive circuitry, through targeted brain stimulation. Previous studies have demonstrated that a single session of 10 Hz transcranial magnetic stimulation (TMS) over the dlPFC can lead to a decrease in craving for alcohol, nicotine, and cocaine. Our laboratory has demonstrated that a single session of continuous theta burst (cTBS) TMS over the mPFC can also decrease craving, as well as the brain response to drug cues in cocaine users (Hanlon et al, in review) and alcohol users (see Significance). The overarching goal of this proposal is to determine which of these two TMS strategies - amplifying dlPFC activity or inhibiting mPFC activity - is more efficacious in decreasing alcohol craving and the brain response to cues. This will provide an evidence-based foundation for cortical target selection in future TMS clinical trials - an innovative treatment strategy for AUD patients.

As a recent FDA-approved treatment for depression, there is a growing interest in investigating TMS as a treatment for drug and alcohol use disorders. By changing the frequency and pattern of stimulation, it is possible to induce a long-term potentiation (LTP) or long-term depression (LTD) of activity in the cortical area stimulated as well in its monosynaptic targets. To date, nearly all published reports of brain stimulation as a tool for decreasing craving have focused on applying LTP-like stimulation (typically 10 Hz) to the dlPFC, thereby strengthening executive control circuitry. An alternative approach is to apply LTD-like TMS (such as cTBS) to the mPFC, thereby weakening limbic drive circuitry (which is engaged during craving). A sham TMS-controlled crossover study of 12 heavy alcohol users in our lab indicated that a single dose of mPFC cTBS decreases self-reported craving and the BOLD response to alcohol cues in the mPFC and striatum (limbic regions involved in craving). Using MR spectroscopy, we further demonstrated that cTBS-reduced the glutamine concentration in the mPFC, which may be related to the decrease in BOLD signal and functional connectivity with this region. Before moving forward with large and expensive multisite clinical trials, it is important to determine which cortical target (mPFC vs dlPFC) is likely to have a greater effect on the brain response to alcohol cues (Aim 1), and which will have a greater effect on self-reported craving (Aim 2) -a major factor contributing to relapse and sustained heavy drinking among individuals with AUDs. In this three-visit crossover design, a cohort of non-treatment seeking AUD individuals will receive sham, mPFC, or dlPFC TMS at each visit followed by alcohol-cue induced BOLD imaging and MR Spectroscopy. We will determine whether LTD-like mPFC TMS is more effective than LTP-like dlPFC TMS in:

Aim 1: Reducing alcohol cue-elicited brain activity in limbic circuitry. Participants will be exposed to our well-established fMRI alcohol cue paradigm. We will measure the percent BOLD signal change within a network of limbic regions typically activated by alcohol cues (e.g. mPFC, ACC, striatum) (Schacht et al., 2014), as well as functional connectivity between these regions (using psychophysiologic interactions). We will test the hypotheses that 1) both LTD-like stimulation to the mPFC (via cTBS) and LTP-like stimulation to the dlPFC (via 10Hz TMS) will significantly decrease alcohol cue-induced activation of limbic circuitry compared to sham stimulation and 2) this attenuating effect will be more robust when stimulation is targeted at the mPFC directly with cTBS stimulation (rather than indirectly via 10 Hz dlPFC stimulation).

Aim 2: Reducing self-reported alcohol craving. Using intermittent self-reported assessments of the desire to drink alcohol throughout the experimental sessions (before, during, and at several time points after the TMS treatment), we will test the hypothesis that LTD-like stimulation to the mPFC (via cTBS) will decrease self-reported alcohol craving more than will LTP-like stimulation to the dlPFC (via 10Hz TMS).

Finally, to develop a comprehensive and evidence-based foundation for future clinical trials, we will also explore the effects of these innovative brain stimulation treatment strategies on neurochemistry:

Exploratory Aim 3: Regional neurochemistry. Through MR Spectroscopy, we will test the hypothesis that the effects of TMS on the outcomes of Aim 1 & 2 are mediated by changes in mPFC excitatory/inhibitory neurochemical balance (i.e., changes in glutamate, glutamine, GABA concentrations).

ELIGIBILITY:
Inclusion Criteria: Age 21-40; Current alcohol use greater than 20 standard drinks per week; Current DSM-5 Alcohol Use Disorder diagnosis, including the loss of control item; Currently not engaged in, and do not want treatment for, alcohol related problems; Able to read and understand questionnaires and informed consent; Lives within 50 miles of the study site. Exclusion Criteria: [These are listed in greater detail in the CIA Core] Any current DSM-5 Axis I diagnosis except Alcohol or Nicotine Use Disorder; Current use of any psychoactive substance except nicotine and marijuana or medication as evidenced by self-report or urine drug screen; History of head trauma or epilepsy; Current suicidal or homicidal ideation; Presence of ferrous metal in the body, as evidenced by metal screening and self-report; Severe claustrophobia or extreme obesity that preclude placement in the MRI scanner. For female participants, pregnancy, as evidenced by a urine pregnancy test administered on the day of the scanning session.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2016-01; Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Percent signal change in the MPFC | immediately after the treatment
Percent signal change in the DLPFC | immediately after the treatment
Change in craving score | immediately after the treatment

SECONDARY OUTCOMES:
Change in glutmate concentration | immediately after the treatment
Change in GABA concentration | immediately after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: James Prisciandaro, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the National Institute of Health Neuroimaging Biorepository at the completion of the study

REFERENCES:
- [Background] Sinha R. New findings on biological factors predicting addiction relapse vulnerability. Curr Psychiatry Rep. 2011 Oct;13(5):398-405. doi: 10.1007/s11920-011-0224-0. PMID 21792580
- [Background] Kalivas PW, Volkow ND. The neural basis of addiction: a pathology of motivation and choice. Am J Psychiatry. 2005 Aug;162(8):1403-13. doi: 10.1176/appi.ajp.162.8.1403. PMID 16055761
- [Background] Sinha R, Catapano D, O'Malley S. Stress-induced craving and stress response in cocaine dependent individuals. Psychopharmacology (Berl). 1999 Mar;142(4):343-51. doi: 10.1007/s002130050898. PMID 10229058
- [Background] Lee JL, Milton AL, Everitt BJ. Cue-induced cocaine seeking and relapse are reduced by disruption of drug memory reconsolidation. J Neurosci. 2006 May 31;26(22):5881-7. doi: 10.1523/JNEUROSCI.0323-06.2006. PMID 16738229
- [Background] Volkow ND, Wang GJ, Fowler JS, Tomasi D. Addiction circuitry in the human brain. Annu Rev Pharmacol Toxicol. 2012;52:321-36. doi: 10.1146/annurev-pharmtox-010611-134625. Epub 2011 Sep 27. PMID 21961707
- [Background] Bolla K, Ernst M, Kiehl K, Mouratidis M, Eldreth D, Contoreggi C, Matochik J, Kurian V, Cadet J, Kimes A, Funderburk F, London E. Prefrontal cortical dysfunction in abstinent cocaine abusers. J Neuropsychiatry Clin Neurosci. 2004 Fall;16(4):456-64. doi: 10.1176/jnp.16.4.456. PMID 15616172
- [Background] Bolla KI, Eldreth DA, London ED, Kiehl KA, Mouratidis M, Contoreggi C, Matochik JA, Kurian V, Cadet JL, Kimes AS, Funderburk FR, Ernst M. Orbitofrontal cortex dysfunction in abstinent cocaine abusers performing a decision-making task. Neuroimage. 2003 Jul;19(3):1085-94. doi: 10.1016/s1053-8119(03)00113-7. PMID 12880834
- [Background] Hanlon CA, Wesley MJ, Stapleton JR, Laurienti PJ, Porrino LJ. The association between frontal-striatal connectivity and sensorimotor control in cocaine users. Drug Alcohol Depend. 2011 Jun 1;115(3):240-3. doi: 10.1016/j.drugalcdep.2010.11.008. Epub 2010 Dec 28. PMID 21193273
- [Background] Gu H, Salmeron BJ, Ross TJ, Geng X, Zhan W, Stein EA, Yang Y. Mesocorticolimbic circuits are impaired in chronic cocaine users as demonstrated by resting-state functional connectivity. Neuroimage. 2010 Nov 1;53(2):593-601. doi: 10.1016/j.neuroimage.2010.06.066. Epub 2010 Jul 11. PMID 20603217
- [Background] Bear MF, Malenka RC. Synaptic plasticity: LTP and LTD. Curr Opin Neurobiol. 1994 Jun;4(3):389-99. doi: 10.1016/0959-4388(94)90101-5. PMID 7919934
- [Background] Malenka RC, Bear MF. LTP and LTD: an embarrassment of riches. Neuron. 2004 Sep 30;44(1):5-21. doi: 10.1016/j.neuron.2004.09.012. PMID 15450156
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Di Lazzaro V, Pilato F, Saturno E, Oliviero A, Dileone M, Mazzone P, Insola A, Tonali PA, Ranieri F, Huang YZ, Rothwell JC. Theta-burst repetitive transcranial magnetic stimulation suppresses specific excitatory circuits in the human motor cortex. J Physiol. 2005 Jun 15;565(Pt 3):945-50. doi: 10.1113/jphysiol.2005.087288. Epub 2005 Apr 21. PMID 15845575
- [Background] Verbruggen F, Aron AR, Stevens MA, Chambers CD. Theta burst stimulation dissociates attention and action updating in human inferior frontal cortex. Proc Natl Acad Sci U S A. 2010 Aug 3;107(31):13966-71. doi: 10.1073/pnas.1001957107. Epub 2010 Jul 14. PMID 20631303
- [Background] Cho SS, Ko JH, Pellecchia G, Van Eimeren T, Cilia R, Strafella AP. Continuous theta burst stimulation of right dorsolateral prefrontal cortex induces changes in impulsivity level. Brain Stimul. 2010 Jul;3(3):170-6. doi: 10.1016/j.brs.2009.10.002. Epub 2009 Oct 31. PMID 20633446
- [Background] Jacobson L, Javitt DC, Lavidor M. Activation of inhibition: diminishing impulsive behavior by direct current stimulation over the inferior frontal gyrus. J Cogn Neurosci. 2011 Nov;23(11):3380-7. doi: 10.1162/jocn_a_00020. Epub 2011 Mar 31. PMID 21452949
- [Background] Camprodon JA, Martinez-Raga J, Alonso-Alonso M, Shih MC, Pascual-Leone A. One session of high frequency repetitive transcranial magnetic stimulation (rTMS) to the right prefrontal cortex transiently reduces cocaine craving. Drug Alcohol Depend. 2007 Jan 5;86(1):91-4. doi: 10.1016/j.drugalcdep.2006.06.002. Epub 2006 Sep 12. PMID 16971058
- [Background] Politi E, Fauci E, Santoro A, Smeraldi E. Daily sessions of transcranial magnetic stimulation to the left prefrontal cortex gradually reduce cocaine craving. Am J Addict. 2008 Jul-Aug;17(4):345-6. doi: 10.1080/10550490802139283. No abstract available. PMID 18612892
- [Background] Barr MS, Fitzgerald PB, Farzan F, George TP, Daskalakis ZJ. Transcranial magnetic stimulation to understand the pathophysiology and treatment of substance use disorders. Curr Drug Abuse Rev. 2008 Nov;1(3):328-39. doi: 10.2174/1874473710801030328. PMID 19630729
- [Background] Wing VC, Barr MS, Wass CE, Lipsman N, Lozano AM, Daskalakis ZJ, George TP. Brain stimulation methods to treat tobacco addiction. Brain Stimul. 2013 May;6(3):221-30. doi: 10.1016/j.brs.2012.06.008. Epub 2012 Jul 9. PMID 22809824
- [Background] Hanlon CA, Canterberry M, Taylor JJ, DeVries W, Li X, Brown TR, George MS. Probing the frontostriatal loops involved in executive and limbic processing via interleaved TMS and functional MRI at two prefrontal locations: a pilot study. PLoS One. 2013 Jul 9;8(7):e67917. doi: 10.1371/journal.pone.0067917. Print 2013. PMID 23874466
- [Background] Bestmann S, Baudewig J, Siebner HR, Rothwell JC, Frahm J. Functional MRI of the immediate impact of transcranial magnetic stimulation on cortical and subcortical motor circuits. Eur J Neurosci. 2004 Apr;19(7):1950-62. doi: 10.1111/j.1460-9568.2004.03277.x. PMID 15078569
- [Background] Bohning DE, Shastri A, Lomarev MP, Lorberbaum JP, Nahas Z, George MS. BOLD-fMRI response vs. transcranial magnetic stimulation (TMS) pulse-train length: testing for linearity. J Magn Reson Imaging. 2003 Mar;17(3):279-90. doi: 10.1002/jmri.10271. PMID 12594717
- [Background] Fox MD, Buckner RL, White MP, Greicius MD, Pascual-Leone A. Efficacy of transcranial magnetic stimulation targets for depression is related to intrinsic functional connectivity with the subgenual cingulate. Biol Psychiatry. 2012 Oct 1;72(7):595-603. doi: 10.1016/j.biopsych.2012.04.028. Epub 2012 Jun 1. PMID 22658708
- [Background] Vernet M, Bashir S, Yoo WK, Oberman L, Mizrahi I, Ifert-Miller F, Beck CJ, Pascual-Leone A. Reproducibility of the effects of theta burst stimulation on motor cortical plasticity in healthy participants. Clin Neurophysiol. 2014 Feb;125(2):320-6. doi: 10.1016/j.clinph.2013.07.004. Epub 2013 Aug 7. PMID 23932365
- [Background] Wilcox CE, Teshiba TM, Merideth F, Ling J, Mayer AR. Enhanced cue reactivity and fronto-striatal functional connectivity in cocaine use disorders. Drug Alcohol Depend. 2011 May 1;115(1-2):137-44. doi: 10.1016/j.drugalcdep.2011.01.009. Epub 2011 Apr 3. PMID 21466926
- [Background] Prisciandaro JJ, McRae-Clark AL, Myrick H, Henderson S, Brady KT. Brain activation to cocaine cues and motivation/treatment status. Addict Biol. 2014 Mar;19(2):240-9. doi: 10.1111/j.1369-1600.2012.00446.x. Epub 2012 Mar 28. PMID 22458561
- [Background] Borckardt JJ, Nahas Z, Koola J, George MS. Estimating resting motor thresholds in transcranial magnetic stimulation research and practice: a computer simulation evaluation of best methods. J ECT. 2006 Sep;22(3):169-75. doi: 10.1097/01.yct.0000235923.52741.72. PMID 16957531